CLINICAL TRIAL: NCT05570201
Title: Effects of Planned Training and Music Listened to Before a Cesarean Section on Surgical Fear, Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sukran Ertekin Pinar, Assoc. Prof.Dr., Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TRSİVAS 01
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Cesarean Section
Keywords: Anxiety and depression; fear of surgery; listening to music; planned training; cesarean section
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): By visiting the women who met the research criteria, the purpose of the study was explained and their written informed consent was obtained. This study was conducted in two sessions using pre- and post-tests. The Personal Information Form, the SFQ, and the HADS were filled out using the face-to-face interview method by the researcher for the women included in the music and training on the day of their hospitalization, which lasted for 30-45 minutes.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Control group — No intervention was applied to the women in the control group, only the questionnaires (pre-test, post-test) were filled out. Filling the questionnaires lasted 10-15 minutes on average in all groups

SUMMARY:
This research was conducted to determine the effect of training and listening to music before a cesarean section on the surgical fear, anxiety and depression

DETAILED DESCRIPTION:
The sample of the experimental study consisted of 120 pregnant women (music: 40, training: 40, control: 40). The data were collected using the Personal Information Form, Surgical Fear Questionnaire, and the Hospital Anxiety and Depression Scale. After the training and listening to music applications, statistically significant differences were found between the music, training, and the control groups in terms of the short-term, long-term sub-scale scores and the overall score of the Surgical Fear Questionnaire, and the anxiety sub-scale scores of the Hospital Anxiety and Depression Scale (p < .05). Listening to music before the cesarean section was effective in reducing women's short-term and general surgical fears, and the training was also effective in reducing their short-term, long-term, and general surgical fears and anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Women who were hospitalized for planned cesarean section,
* Having the first pregnancy,
* Between the ages 19 and 35,
* Who had no diagnosis of a physical or mental disease,
* Who had no physical illness in her baby

Exclusion Criteria:

-

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Likert type scale | 15 months
  The scale is an 11-point Likert type scale, consisting of 8 items, scored between 0 and 10 points each. The scale consists of two sub-scales, consisting of 4 items each, measuring short-term fears and long-term fears related to the source of fear. The items in the scale are evaluated as "0:I am not afraid at all" to "10:I am very afraid".

SECONDARY OUTCOMES:
Anxiety and Depression sub-scale | 15 months
  It is used for diagnosing anxiety and depression in a short time and determining the risk group. It's a 4-point Likert-type scale consisting of 14 items in total. There are 7 items in the Anxiety and Depression sub-scale, and they are scored in the range of 0-3 points. The lowest and highest scores that can be taken in the sub-scales are 0 and 21, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: sukran Ertekin Pınar, Principal Investigator — Cumhuriyet Universty
Locations (1):
- Sukran Ertekin Pınar, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Baert IA, Lluch E, Mulder T, Nijs J, Noten S, Meeus M. Does pre-surgical central modulation of pain influence outcome after total knee replacement? A systematic review. Osteoarthritis Cartilage. 2016 Feb;24(2):213-23. doi: 10.1016/j.joca.2015.09.002. Epub 2015 Sep 14. PMID 26382109
- [Background] Bastani F, Hidarnia A, Montgomery KS, Aguilar-Vafaei ME, Kazemnejad A. Does relaxation education in anxious primigravid Iranian women influence adverse pregnancy outcomes?: a randomized controlled trial. J Perinat Neonatal Nurs. 2006 Apr-Jun;20(2):138-46. doi: 10.1097/00005237-200604000-00007. PMID 16714913
- [Background] Cooke M, Chaboyer W, Schluter P, Hiratos M. The effect of music on preoperative anxiety in day surgery. J Adv Nurs. 2005 Oct;52(1):47-55. doi: 10.1111/j.1365-2648.2005.03563.x. PMID 16149980
- [Background] Eslami J, Hatami N, Amiri A, Akbarzadeh M. The potential beneficial effects of education and familiarity with cesarean section procedure and the operating room environment on promotion of anxiety and pain intensity: A randomized controlled clinical trial. J Educ Health Promot. 2020 Sep 28;9:240. doi: 10.4103/jehp.jehp_31_20. eCollection 2020. PMID 33209932
- [Background] Hepp P, Hagenbeck C, Gilles J, Wolf OT, Goertz W, Janni W, Balan P, Fleisch M, Fehm T, Schaal NK. Effects of music intervention during caesarean delivery on anxiety and stress of the mother a controlled, randomised study. BMC Pregnancy Childbirth. 2018 Nov 3;18(1):435. doi: 10.1186/s12884-018-2069-6. PMID 30390639
- [Background] Shabel'nik DIa, Grinchishin SA. [Polychlorpinene poisoning]. Sud Med Ekspert. 1969 Jul-Sep;12(3):47-8. No abstract available. Russian. PMID 5382598
- [Background] Kiyohara LY, Kayano LK, Oliveira LM, Yamamoto MU, Inagaki MM, Ogawa NY, Gonzales PE, Mandelbaum R, Okubo ST, Watanuki T, Vieira JE. Surgery information reduces anxiety in the pre-operative period. Rev Hosp Clin Fac Med Sao Paulo. 2004 Apr;59(2):51-6. doi: 10.1590/s0041-87812004000200001. Epub 2004 Apr 26. PMID 15122417
- [Background] Liu YH, Chang MY, Chen CH. Effects of music therapy on labour pain and anxiety in Taiwanese first-time mothers. J Clin Nurs. 2010 Apr;19(7-8):1065-72. doi: 10.1111/j.1365-2702.2009.03028.x. PMID 20492051
- [Background] Moutzouri M, Gleeson N, Billis E, Tsepis E, Panoutsopoulou I, Gliatis J. The effect of total knee arthroplasty on patients' balance and incidence of falls: a systematic review. Knee Surg Sports Traumatol Arthrosc. 2017 Nov;25(11):3439-3451. doi: 10.1007/s00167-016-4355-z. Epub 2016 Oct 19. PMID 27761627
- [Background] Ramesh C, Nayak BS, Pai VB, Patil NT, George A, George LS, Devi ES. Effect of Preoperative Education on Postoperative Outcomes Among Patients Undergoing Cardiac Surgery: A Systematic Review and Meta-Analysis. J Perianesth Nurs. 2017 Dec;32(6):518-529.e2. doi: 10.1016/j.jopan.2016.11.011. Epub 2017 Apr 13. PMID 29157759
- [Background] Ribeiro MKA, Alcantara-Silva TRM, Oliveira JCM, Paula TC, Dutra JBR, Pedrino GR, Simoes K, Sousa RB, Rebelo ACS. Music therapy intervention in cardiac autonomic modulation, anxiety, and depression in mothers of preterms: randomized controlled trial. BMC Psychol. 2018 Dec 13;6(1):57. doi: 10.1186/s40359-018-0271-y. PMID 30545420
- [Background] Ruhaiyem ME, Alshehri AA, Saade M, Shoabi TA, Zahoor H, Tawfeeq NA. Fear of going under general anesthesia: A cross-sectional study. Saudi J Anaesth. 2016 Jul-Sep;10(3):317-21. doi: 10.4103/1658-354X.179094. PMID 27375388
- [Background] Shimada BMO, Santos MDSOMD, Cabral MA, Silva VO, Vagetti GC. Interventions among Pregnant Women in the Field of Music Therapy: A Systematic Review. Rev Bras Ginecol Obstet. 2021 May;43(5):403-413. doi: 10.1055/s-0041-1731924. Epub 2021 Jun 28. PMID 34182584
- [Background] Sun Y, Huang K, Hu Y, Yan S, Xu Y, Zhu P, Tao F. Pregnancy-specific anxiety and elective cesarean section in primiparas: A cohort study in China. PLoS One. 2019 May 15;14(5):e0216870. doi: 10.1371/journal.pone.0216870. eCollection 2019. PMID 31091276
- [Background] Theunissen M, Peters ML, Schouten EG, Fiddelers AA, Willemsen MG, Pinto PR, Gramke HF, Marcus MA. Validation of the surgical fear questionnaire in adult patients waiting for elective surgery. PLoS One. 2014 Jun 24;9(6):e100225. doi: 10.1371/journal.pone.0100225. eCollection 2014. PMID 24960025
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Bagdigen M, Karaman Ozlu Z. Validation of the Turkish Version of the Surgical Fear Questionnaire. J Perianesth Nurs. 2018 Oct;33(5):708-714. doi: 10.1016/j.jopan.2017.05.007. Epub 2017 Sep 21. PMID 30236578
- See also: Relationship Between Perceived Social Support and Anxiety Before and After Cesarean in the Pregnant Women — http://biomedres.us/fulltexts/BJSTR.MS.ID.005528.php
- See also: Impact of Face-to-Face Educational Outreach Plus Printed Materials on Preoperative Anxiety level in Iranian Parturient Undergoing Elective Cesarean Section Delivery — https://aacc.tums.ac.ir/index.php/aacc/article/view/214
- See also: Effect of Education and Musical Therapy Given During Labor on the Process of Birth in Induced Primipara Pregnant Women — https://valleyinternational.net/index.php/ijmsci/article/view/731